CLINICAL TRIAL: NCT00285181
Title: Effects of Statins on Pro- and Antioxidant Status : Link With Statin-Associated Myopathy. A Randomized, Placebo-Controlled, Double-Blind Study.
Brief Title: Effects of Statins on Pro- and Antioxidant Status : Link With Statin-Associated Myopathy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UF7808
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2007-08-09 (Estimated); Status verified 2007-08

CONDITIONS: Healthy
Keywords: persons
MeSH Terms: interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Simvastatin

SUMMARY:
To evaluate the effects of a 8-week treatment with 80 mg/day simvastatin on prooxidant and antioxidant status at rest and after exercise, on mitochondrial respiration and calcium release in skeletal muscle, and on aérobic aptitude in 24 healthy male subjects.

DETAILED DESCRIPTION:
Day 1 : baseline oxidative status, lipid profile, exercice test, start of randomized treatment Day 53 : muscular biopsy Day 57 : follow-up oxidative status, lipid profile, exercice test, end of treatment

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.0 and 25.00

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2005-11; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Blood antioxidant status before treatment and after treatment.
Lipid and protein peroxidation indexes before treatment and after treatment.
In vitro mitochondrial respiration, enzymatic activities and calcium release parameters before treatment and after treatment.

SECONDARY OUTCOMES:
Blood lipids before treatment and after treatment
LDL composition before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre PETIT, MD-PhD, Principal Investigator — Centre d'Investigation Clinique
Locations (1):
- Centre d'Investigation Clinique, Montpellier, France